CLINICAL TRIAL: NCT01531751
Title: An Open Label Phase II Trial of Free Light Chain Removal by Extended High Cut-Off Hemodialysis in Patients With Advanced Cardiac AL Amyloidosis and End-Stage Renal Disease.
Brief Title: High Cut-off Hemodialysis in Patients With Advanced Cardiac AL Amyloidosis and End Stage Renal Disease
Acronym: DIACAL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giampaolo Merlini, Director, Amyloidosis Research and Treatment Center, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-005-IT
Record Dates: First submitted 2012-01-11; First posted 2012-02-13 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Primary Amyloidosis of Light Chain Type
Keywords: HCO-HD; survival; cardiac biomarkers; AL amyloidosis; Light Chain Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Cut-off Hemodialysis (Experimental)
  Interventions: Device: High Cut-off Hemodialysis; Drug: Chemotherapy

INTERVENTIONS:
Device: High Cut-off Hemodialysis — During dialysis the patients will undergo the first cycle of chemotherapy according to the current standard of care for subjects with advanced cardiac AL amyloidosis. Measurements of FLC and cardiac biomarkers will be done before and after each dialysis session. High cutoff HD will be continued during the first chemotherapy cycle. After the first cycle the end-of-treatment evaluation will take place.
  Other Names: Theralite
Drug: Chemotherapy — Chemotherapy will be based on alchilators, proteasome inhibitors, steroids, IMiDs.

SUMMARY:
The aim of the study is to assess survival of patients with advanced cardiac AL amyloidosis treated with high cut-off hemodialysis (HCO-HD) combined with chemotherapy.

DETAILED DESCRIPTION:
This will be a single-center phase II open label trial. Subjects with advanced cardiac AL amyloidosis and end-stage renal disease will undergo HCO-HD while receiving chemotherapy for their plasma cell dyscrasia according to the current standards of care.

After giving written informed consent, the patients will be evaluated for eligibility. Briefly, the subjects with a biopsy-proven diagnosis of AL amyloidosis who are cardiac stage 3 based on NT-proBNP (> 332 ng/L) and cTnI (> 100 ng/L) and whose estimated glomerular filtration rate (eGFR) is < 15 mL/min per 1.73 m2 will be eligible for the study. Patients with non-AL (e.g. familial and senile) amyloidosis will be excluded, as well as subjects who have less than 100 mg/L circulating amyloidogenic FLC. Sixteen patients will be enrolled.

The study includes 3 periods: screening, treatment followed by the end-of-treatment evaluation and follow-up. During dialysis the patients will undergo the first cycle of chemotherapy according to the current standard of care for subjects with advanced cardiac AL amyloidosis. Measurements of FLC and cardiac biomarkers will be done before and after each dialysis session. High cutoff HD will be continued during the first chemotherapy cycle. After the first cycle the end-of-treatment evaluation will take place. Follow-up evaluations will be performed after the end of each subsequent chemotherapy cycle and every 2 months after chemotherapy discontinuation for 1 year or until disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AL amyloidosis.
* Age ≥ 18 years.
* Evidence of a monoclonal light chain in serum and/or urine by positive immunofixation and abnormal FLC κ/λ ratio.
* Evidence of cardiac involvement at echocardiography (mean left ventricular wall thickness > 12 mm in the absence of other causes).
* Cardiac stage III (both NT-proBNP > 332 ng/L and cTnI > 100 ng/L).
* Estimated GFR < 15 mL/min per 1.73 m2 or requiring dialysis.
* NYHA class III or IV.
* Initiation of chemotherapy for AL amyloidosis scheduled between day 3 and day 8 after first HCO-HD session.

Exclusion Criteria:

* Non-AL (e.g. familial, senile) amyloidosis.
* Concomitant non-amyloid related clinically significant cardiac diseases.
* Involved (amyloidogenic) FLC < 100 mg/L.
* Inability to undergo chemotherapy for AL amyloidosis.
* Uncontrolled infection.
* Inability to give informed consent.
* Previous or ongoing psychiatric illness (excluding reactive depression).
* Pregnant or nursing women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Survival | 6 months
  The primary objective will be to assess survival of patients with advanced cardiac AL amyloidosis treated with HCO-HD combined with chemotherapy.

SECONDARY OUTCOMES:
tolerability of the experimental device | 1 month
  Secondary objectives will be to assess the feasibility and tolerability of HCO-HD in patients with advanced cardiac AL amyloidosis, the efficiency of HCO-HD plus chemotherapy in reducing amyloidogenic FLC in this setting, and the ability of this approach to promote improvement of cardiac dysfunction as assessed by biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro per lo Studio e la Cura delle Amiloidosi Sistemiche - Fondazione IRCCS Policlinico S.Matteo, Pavia, Italy

REFERENCES:
- [Background] Hutchison CA, Cockwell P, Reid S, Chandler K, Mead GP, Harrison J, Hattersley J, Evans ND, Chappell MJ, Cook M, Goehl H, Storr M, Bradwell AR. Efficient removal of immunoglobulin free light chains by hemodialysis for multiple myeloma: in vitro and in vivo studies. J Am Soc Nephrol. 2007 Mar;18(3):886-95. doi: 10.1681/ASN.2006080821. Epub 2007 Jan 17. PMID 17229909
- See also: Related Info — http://www.amiloidosi.it/